CLINICAL TRIAL: NCT02798653
Title: Comparison of Different Methods for Luteal Phase Support in IVF / ICSI Cycles With Antagonist Protocol in Women With Poor Ovarian Response
Brief Title: Evaluation of Different Luteal Phase Support Methods in Patients With Poor Ovarian Response
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-024
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2016-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Choriomon® (Experimental): subjects receive 1,500 IU of hCG (Choriomon®; IBSA) intramuscular (IM) on the embryos transfer (ET) day, as well as 4 days after the embryos transfer for luteal support
  Interventions: Drug: Choriomon® injection
- Choriomon®+Endometrin ® (Experimental): patients will receive 1,500 IU of hCG (Choriomon®; IBSA) (IM) on the ET day, as well as 3 and 6 days after the transfer along with Endometrin ® vaginal tablets (Ferring Pharmaceuticals Ltd., Germany) 100 mg twice daily for luteal support from the day of oocyte pickup to the day of the pregnancy test.
  Interventions: Drug: Choriomon® injection+Endometrin ®
- Endometrin ® (Experimental): patients will receive only Endometrin ® vaginal tablets (Ferring Pharmaceuticals Ltd., Germany) 100 mg twice daily for luteal support from the day of oocyte pickup to the day of the pregnancy test.
  Interventions: Drug: Endometrin ® vaginal tablets

INTERVENTIONS:
Drug: Choriomon® injection — Intramuscular injection of 1,500 IU of hCG (Choriomon®; IBSA) on the embryos transfer (ET) day, as well as 4 days after the embryos transfer for luteal support
  Arms: Choriomon®
Drug: Choriomon® injection+Endometrin ® — Intramuscular injection of 1,500 IU of hCG (Choriomon®; IBSA) on the ET day, as well as 3 and 6 days after the transfer along with Endometrin ® vaginal tablets (Ferring Pharmaceuticals Ltd., Germany) 100 mg twice daily for luteal support from the day of oocyte pickup to the day of the pregnancy test.
  Arms: Choriomon®+Endometrin ®
Drug: Endometrin ® vaginal tablets — Endometrin ® vaginal tablets (Ferring Pharmaceuticals Ltd., Germany) 100 mg twice daily for luteal support from the day of oocyte pickup to the day of the pregnancy test.
  Arms: Endometrin ®

SUMMARY:
This study is a randomized clinical trial to investigate the efficacy of different luteal phase support methods in patients with poor ovarian response undergoing IVF and intracytoplasmic sperm injection (ICSI) cycles.

The study protocol is approved by the Ethics Committee (Institutional Review Board) of Royan institute. The study is conducted according to the Declaration of Helsinki for medical research. All participants provide informed consent after counseling for infertility treatments and routine IVF/ICSI programs.

DETAILED DESCRIPTION:
All the patients who diagnose as poor ovarian responders (POR) based on the Bologna criteria are eligible for participation in this study. In order to define the poor response in IVF, at least two of the following three features must be present: (i) advanced maternal age or any other risk factor for POR; (ii) a previous POR; and (iii) an abnormal ovarian reserve test (ORT). Two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ORT.

The ovarian stimulation is performed with antagonist protocol with E2 priming for all eligible patients. All women receive estrogen priming (E2 tablet) starting a week after LH surge until menses. Controlled ovarian stimulation is started on day 2 of menstrual cycle with 225 IU recombinant FSH (Gonal-F®; Serono Laboratories Ltd., Geneva, Switzerland) and 75 IU hMG (Menopur®; Ferring). The doses of gonadotropins were adjusted as ovarian response in the ultrasound monitoring. Gonadotropin releasing hormone (GnRH) antagonist (Cetrorelix acetate 0.25 mg; Cetrotide ®, USAN) is administrated to prevent premature ovulation when the lead follicle measured ≥ 12 mm and was continued until the hCG trigger. Final oocyte triggering will be done with 10000 IU of hCG (Choriomon®; IBSA). If there were or more dominant follicles, oocytes retrieval will be done under transvaginal ultrasound guidance 32-34 hours after hCG administration. Intracytoplasmic sperm injection will be performed for all metaphase II oocytes. Embryo transfer will be done under ultrasound guidance on day 3 for all patients.

On the day of oocyte pickup, patients are allocated randomly (by the blocked randomization method) into three groups to receive three different luteal support protocols and they remained on the same allocation throughout the study. Group 1, subjects receive 1,500 IU of hCG IM on the embryos transfer (ET) day, as well as 4 days after the embryos transfer. Group 2: patients will receive 1,500 IU of hCG IM on the ET day, as well as 3 and 6 days after the transfer along with Endometrin ® vaginal tablets (Ferring Pharmaceuticals Ltd., Germany) 100 mg twice daily. Group 3, patients will receive only Endometrin ® vaginal tablets (Ferring Pharmaceuticals Ltd., Germany) 100 mg twice daily for luteal support from the day of oocyte pickup to the day of the pregnancy test. The vaginal progesterone is continued in all patients who become pregnant in all three groups until the 12th week of pregnancy. The serum ß-hCG level is checked 2 weeks after ET to confirm positive pregnancy test. Clinical pregnancies are detected with the confirmation of positive fetal heart activities by transvaginal sonography. The implantation rate is considered as the proportion of number of observed intrauterine gestational sac to number of transferred embryos. Multiple pregnancies are defined as two or more gestational sacs in the uterine cavity. Miscarriage is defined as a loss of a clinical pregnancy before the 12th week of gestation.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of poor ovarian response (POR), according to Bologna criteria:

the patients have at least two of the following criteria:

* age over 40 years;
* a history of ovarian surgery;
* previous treatment using conventional protocols that yielded less than three oocytes;
* antral follicle count of less than 5 on menstrual cycle day 2-3; and basal serum FSH concentration between 10 and 19 IU/l or serum anti-Müllerian hormone level less than 1 ng/ml.

Exclusion Criteria:

1- Female age over 45 years old 2- Ovarian failure including basal FSH above 20 IU/l or no antral follicle by ultrasound examination 3- Severe male factor (Azoospermia) 4- Endometriosis diagnosis and the presence of hydrosalpinges 5- Uterine factor (polyps, myoma and previous myomectomy, …) 6- Patients with cardiovascular disease and/or uncontrolled systemic or endocrine diseases 7- Patients with repeated implantation failures and repeated miscarriages. 8- Female smokers

-

Ages: 40 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks
  Evaluation the clinical pregnancy rate at least 4 weeks after embryo transfer.

SECONDARY OUTCOMES:
Implantation rate | 4 weeks
  Evaluation the implantation rate at least 4 weeks after embryo transfer
chemical pregnancy rates | 2 weeks
  Evaluation of chemical pregnancy rates 2 weeks after embryo transfer
miscarriage rate | 12 weeks
  Evaluation of miscarriage rate 12 weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, p, Study Chair — Head of Royan Institute; Tahere Madani, MD, Study Director — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Fariba Ramezani, MD, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Arezoo Arabipour, M.S.c, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Madani T, Arabipoor A, Ramezanali F, Khodabakhshi S, Zolfaghary Z. The Effects of Three Methods of Luteal Phase Support on Pregnancy Outcomes in Poor Ovarian Responders: A Randomized Clinical Trial. Int J Fertil Steril. 2025 Jan 5;19(1):10-16. doi: 10.22074/ijfs.2024.2007292.1500. PMID 39827385
- See also: Related Info — http://royaninstitute.org